CLINICAL TRIAL: NCT07309562
Title: A Multicenter, Randomized, Open-Label, Active-Controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of Inpegsomatropin Injection, s.c Once a Week, Compared With Recombinant Human Growth Hormone (rhGH) Injection in Children With Short Stature Born Small for Gestational Age（SGA）
Brief Title: The Efficacy and Safety of Inpegsomatropin Injection in Children With Short Stature Born Small for Gestational Age
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEGPESEN-4-2-002
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Small for Gestational Age
Keywords: Inpegsomatropin Injection; Recombinant Human Growth Hormone Injection
MeSH Terms: interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group 1 (Experimental)
  Interventions: Drug: Inpegsomatropin Injection
- Experimental Group 2 (Experimental)
  Interventions: Drug: Inpegsomatropin Injection
- rhGH group (Active Comparator)
  Interventions: Drug: Recombinant Human Growth Hormone Injection

INTERVENTIONS:
Drug: Inpegsomatropin Injection — Inpegsomatropin injection, 140 μg/kg/week, s.c., once weekly, for 52 weeks.
  Arms: Experimental Group 1
Drug: Inpegsomatropin Injection — Inpegsomatropin injection, 280 μg/kg/week, s.c., once weekly, for 52 weeks.
  Arms: Experimental Group 2
Drug: Recombinant Human Growth Hormone Injection — Recombinant human growth hormone injection, 0.033mg/kg/day, s.c.,once daily, for 52 weeks.
  Arms: rhGH group

SUMMARY:
This is a multicenter, randomized, open-label, active-controlled Phase III clinical trial to evaluate the efficacy and safety of Inpegsomatropin injection，once a week，compared with recombinant human growth hormone (rhGH) in children with short stature born small for gestational age (SGA).It plans to enroll 141 children with short stature born small for gestational age (SGA), who will be stratified by gender and age and randomized in a 1:1:1 ratio to either Experimental Group 1, Experimental Group 2, or the Active Control Group. All participants will undergo a screening period (up to 12 weeks), a treatment period (52 weeks), and a post-treatment follow-up period (5 weeks). Safety and efficacy will be comprehensively evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Prepubertal (Tanner stage I) children: boys aged ≥2 and <11 years, and girls aged ≥2 and <10 years at screening.
* Bone age is not more than 1 year advanced or more than 2 years delayed compared to chronological age (i.e., -2 years ≤ bone age - chronological age ≤ 1 year).
* Birth weight and/or length below the 10th percentile for gestational age and sex, according to the reference values in Appendix 1.
* Gestational age at birth ≥28 weeks.
* Height at screening below -2 SD for age and sex, according to the reference values in Appendix 2.
* Body mass index (BMI) between the 5th and 95th percentiles for age and sex, according to the reference values in Appendix 3.
* Peak GH level ≥10.0 ng/mL in at least one prior GH stimulation test.
* No prior systemic growth-promoting therapy (used continuously for ≥1 month), including but not limited to growth hormone, insulin-like growth factor-1 (IGF-1), etc.
* Legal guardian has provided written informed consent. If the participant is ≥8 years old, they must also provide written assent. For participants under 8 years old who are capable of expressing agreement, their assent should be formally documented.

Exclusion Criteria:

* Subjects with closed epiphyses.
* Subjects with other types of growth abnormalities, including confirmed or highly suspected growth hormone deficiency (GHD), Noonan syndrome, Prader-Willi syndrome, Russell-Silver syndrome, Turner syndrome, short stature due to GH receptor deficiency, short stature due to growth plate-related gene abnormalities (e.g., SHOX gene anomalies), growth retardation due to malnutrition, or growth retardation due to hypothyroidism.
* Participation in any other clinical trial with drug or non-drug interventions within 3 months prior to screening.
* Use of inhaled corticosteroids for more than 2 consecutive weeks, or oral/intravenous corticosteroids for more than 1 consecutive week, within 3 months prior to screening.
* Current or long-term requirement for therapies that may affect growth, including but not limited to methylphenidate, sex hormones, gonadotropin-releasing hormone analogs, aromatase inhibitors, anabolic agents, or insulin.
* Abnormal liver or kidney function at screening (ALT > 1.5 times the upper limit of normal [ULN], Cr > ULN).
* Diagnosis of diabetes mellitus, or two consecutive fasting blood glucose measurements ≥ 6.1 mmol/L prior to randomization.
* Chronic infectious diseases which, in the investigator's judgment, may affect study participation (e.g., chronic hepatitis B).
* Systemic chronic diseases, such as chronic kidney disease, severe cardiovascular diseases, or psychiatric/psychological disorders.
* Congenital skeletal dysplasia, scoliosis exceeding 15°, limping gait, or a prior diagnosis of slipped capital femoral epiphysis.
* History of intracranial hypertension.
* Past or current history of malignant tumors, including intracranial tumors.
* Known allergy to growth hormone or any of its excipients.
* Any other condition deemed by the investigator as inappropriate for participation in this clinical trial.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 141 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-05-07 (Estimated)

PRIMARY OUTCOMES:
Growth velocity (HV, cm/year). | Week 52

SECONDARY OUTCOMES:
Change in height standard deviation score from baseline (△HT SDS) | From baseline to all follow-up time points at Week 52
Change in growth velocity from baseline (△HV) | From baseline to all follow-up time points at Week 52
Change in insulin-like growth factor 1 standard deviation score from baseline (△IGF-1 SDS) | From baseline to all follow-up time points at Week 52
Ratio of the change in bone age to the change in chronological age | Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Luo, Ph.D, Principal Investigator — Tongji Hospital
Locations (47):
- China (47):
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing
  - The First Hospital of Jilin University, Changchun
  - Hunan Children's Hospital, Changsha
  - Chengdu Women's and Children's Central Hospital, Chengdu
  - West China Second University Hospital, Sichuan University, Chengdu
  - Children's Hospital of Chongqing Medical University, Chongqing
  - Guangzhou Women and Children's Medical Center, Guangzhou Medical University, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - Hainan Women and Children's Medical Center, Haikou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Heilongjiang Provincial Hospital, Harbin
  - Anhui Children's Hospital, Hefei
  - The Second Affiliated Hospital of Anhui Medical University, Hefei
  - Inner Mongolia People's Hospital, Hohhot
  - Shandong Provincial Hospital, Jinan
  - Affiliated Hospital of Jining Medical University, Jining
  - Jiujiang Maternal and Child Health Hospital, Jiujiang
  - Kunming Children's Hospital, Kunming
  - Gansu Provincial Maternity and Child-care Hospital (Gansu Provincial Central Hospital), Lanzhou
  - Liuzhou People's Hospital, Liuchow
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Jiangxi Provincial Children's Hospital, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Children's Hospital, Nanjing
  - Ningbo Women and Children's Hospital, Ningbo University, Ningbo
  - Qujing Maternal and Child Health Hospital, Qujing
  - Sanya Central Hospital (Hainan Third People's Hospital), Sanya
  - Shanghai Children's Hospital, Shanghai
  - Shanghai Children's Medical Center, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - Children's Hospital of Soochow University, Suzhou
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Wuhan Children's Hospital, Wuhan
  - Wuxi Children's Hospital, Wuxi
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Xiamen Maternal and Child Health Hospital, Xiamen
  - Xuzhou Children's Hospital, Xuzhou
  - Yuncheng Central Hospital, Shanxi Province, Yuncheng
  - Henan Children's Hospital (Zhengzhou Children's Hospital), Zhengzhou
  - Zhuzhou Central Hospital, Zhuzhou

IPD SHARING:
Plan to Share IPD: No